CLINICAL TRIAL: NCT02183675
Title: Pharmacokinetics of Multiple Oral Doses of Telmisartan 80 mg/Amlodipine 5 mg/Hydrochlorothiazide 12.5 mg Fixed-dose Combination Tablet, Telmisartan 80 mg/Hydrochlorothiazide 12.5 mg Fixed-dose Combination Tablet and Telmisartan 80 mg/Amlodipine 5 mg Fixed-dose Combination Tablet at Steady State in Healthy Male Subjects: an Open-label, Randomised, Multiple-dose, Three Treatment, Three-period, Six-sequence Crossover Study
Brief Title: Pharmacokinetics of Different Formulations of Telmisartan, Amlodipine, and Hydrochlorothiazide (HCTZ) in Japanese Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1348.5
Record Dates: First submitted 2014-07-07; First posted 2014-07-08 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
MeSH Terms: interventions — telmisartan amlodipine combination; Telmisartan

ARMS (3):
- T/A/H (Experimental): Telmisartan/Amlodipine/HCTZ fixed-dose combination
  Interventions: Drug: Telmisartan/Amlodipine/HCTZ
- T/A (Active Comparator): Telmisartan/Amlodipine fixed-dose combination
  Interventions: Drug: Telmisartan/Amlodipine
- T/H (Active Comparator): Telmisartan/HCTZ fixed-dose combination
  Interventions: Drug: Telmisartan/HCTZ

INTERVENTIONS:
Drug: Telmisartan/Amlodipine — Telmisartan/Amlodipine fixed-dose combination
  Arms: T/A
Drug: Telmisartan/Amlodipine/HCTZ — Telmisartan/Amlodipine/HCTZ fixed-dose combination
  Arms: T/A/H
Drug: Telmisartan/HCTZ — Telmisartan/HCTZ fixed-dose combination
  Arms: T/H

SUMMARY:
To assess drug drug interaction through pharmacokinetics investigation at steady state of Telmisartan, Amlodipine, and Hydrochlorothiazide (HCTZ) given as three different formulations in healthy Japanese male subjects

ELIGIBILITY:
Inclusion criteria:

* Healthy Japanese male subjects age >=20 and <=35 years; body weight: >=50 kg and <=80 kg; body mass index: >=18.0 and <=25.0 kg/m2
* Without any clinically significant findings and complications on the basis of a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR), body temperature), 12-lead electrocardiograms (ECGs), clinical laboratory tests
* Signed and dated written informed consent prior to admission to the trial in accordance with the Good Clinical Practice (GCP) and the local legislation.

Exclusion criteria:

- Any finding of the medical examination (including BP, PR and ECGs) deviating from normal and of clinical relevance.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1348.5.001 Boehringer Ingelheim Investigational Site, Kanagawa , Yokohama, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, randomised, six-sequence crossover design. Each participant received three treatments each for 10 days. There was no washout period between treatments.
Groups:
- T80-A5-H12.5 / T80-H12.5 / T80-A5: Participants received the three treatments, the treatments were administered orally in the following order:
  * Telmisartan 80mg/Amlodipine 5mg/ hydrochlorothiazide (HCTZ) 12.5mg fixed-dose combination tablet (T80-A5-H12.5)
  * Telmisartan 80mg/ HCTZ 12.5mg fixed-dose combination tablet (T80-H12.5)
  * Telmisartan 80mg/Amlodipine 5mg fixed-dose combination tablet (T80-A5)
- T80-H12.5 / T80-A5 / T80-A5-H12.5: Participants received the three treatments, the treatments were administered orally in the following order:
  * Telmisartan 80mg/HCTZ 12.5mg fixed-dose combination tablet (T80-H12.5)
  * Telmisartan 80mg/Amlodipine 5mg fixed-dose combination tablet (T80-A5)
  * Telmisartan 80mg/Amlodipine 5mg/HCTZ 12.5mg fixed-dose combination tablet (T80-A5-H12.5)
- T80-A5 / T80-A5-H12.5 / T80-H12.5: Participants received the three treatments, the treatments were administered orally in the following order:
  * Telmisartan 80mg/Amlodipine 5mg fixed-dose combination tablet (T80-A5)
  * Telmisartan 80mg/Amlodipine 5mg/HCTZ 12.5mg fixed-dose combination tablet (T80-A5-H12.5)
  * Telmisartan 80mg/HCTZ 12.5mg fixed-dose combination tablet (T80-H12.5)
- T80-A5 / T80-H12.5 / T80-A5-H12.5: Participants received the three treatments, the treatments were administered orally in the following order:
  * Telmisartan 80mg/Amlodipine 5mg fixed-dose combination tablet (T80-A5)
  * Telmisartan 80mg/HCTZ 12.5mg fixed-dose combination tablet (T80-H12.5)
  * Telmisartan 80mg/Amlodipine 5mg/HCTZ 12.5mg fixed-dose combination tablet (T80-A5-H12.5)
- T80-A5-H12.5 / T80-A5 / T80-H12.5: Participants received the three treatments, the treatments were administered orally in the following order:
  * Telmisartan 80mg/Amlodipine 5mg/HCTZ 12.5mg fixed-dose combination tablet (T80-A5-H12.5)
  * Telmisartan 80mg/Amlodipine 5mg fixed-dose combination tablet (T80-A5)
  * Telmisartan 80mg/HCTZ 12.5mg fixed-dose combination tablet (T80-H12.5)
- T80-H12.5 / T80-A5-H12.5 / T80-A5: Participants received the three treatments, the treatments were administered orally in the following order:
  * Telmisartan 80mg/HCTZ 12.5mg fixed-dose combination tablet (T80-H12.5)
  * Telmisartan 80mg/Amlodipine 5mg/HCTZ 12.5mg fixed-dose combination tablet (T80-A5-H12.5)
  * Telmisartan 80mg/Amlodipine 5mg fixed-dose combination tablet (T80-A5)
Period: Treatment Period 1 (10 Days)
Arm/Group | T80-A5-H12.5 / T80-H12.5 / T80-A5 | T80-H12.5 / T80-A5 / T80-A5-H12.5 | T80-A5 / T80-A5-H12.5 / T80-H12.5 | T80-A5 / T80-H12.5 / T80-A5-H12.5 | T80-A5-H12.5 / T80-A5 / T80-H12.5 | T80-H12.5 / T80-A5-H12.5 / T80-A5
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (10 Days)
Arm/Group | T80-A5-H12.5 / T80-H12.5 / T80-A5 | T80-H12.5 / T80-A5 / T80-A5-H12.5 | T80-A5 / T80-A5-H12.5 / T80-H12.5 | T80-A5 / T80-H12.5 / T80-A5-H12.5 | T80-A5-H12.5 / T80-A5 / T80-H12.5 | T80-H12.5 / T80-A5-H12.5 / T80-A5
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 4 (Patients withdrew after completion of treatment period 2 but before beginning of treatment period 3)
Not Completed | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2
Period: Treatment Period 3 (10 Days)
Arm/Group | T80-A5-H12.5 / T80-H12.5 / T80-A5 | T80-H12.5 / T80-A5 / T80-A5-H12.5 | T80-A5 / T80-A5-H12.5 / T80-H12.5 | T80-A5 / T80-H12.5 / T80-A5-H12.5 | T80-A5-H12.5 / T80-A5 / T80-H12.5 | T80-H12.5 / T80-A5-H12.5 / T80-A5
Started | 6 | 6 | 6 | 6 | 6 | 4
Completed | 6 | 6 | 6 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all subjects that were dispensed study drug and were documented to have taken at least one dose of study drug.
Groups:
- T80-A5-H12.5 / T80-H12.5 / T80-A5: Participants received the three treatments, the treatments were administered orally in the following order:
  * Telmisartan 80mg/Amlodipine 5mg/HCTZ 12.5mg fixed-dose combination tablet (T80-A5-H12.5)
  * Telmisartan 80mg/HCTZ 12.5mg fixed-dose combination tablet (T80-H12.5)
  * Telmisartan 80mg/Amlodipine 5mg fixed-dose combination tablet (T80-A5)
- Total: Total of all reporting groups
Arm/Group | T80-A5-H12.5 / T80-H12.5 / T80-A5 | T80-H12.5 / T80-A5 / T80-A5-H12.5 | T80-A5 / T80-A5-H12.5 / T80-H12.5 | T80-A5 / T80-H12.5 / T80-A5-H12.5 | T80-A5-H12.5 / T80-A5 / T80-H12.5 | T80-H12.5 / T80-A5-H12.5 / T80-A5 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.0 (4.9) | 27.3 (5.2) | 27.0 (4.2) | 25.8 (4.1) | 29.5 (5.1) | 29.3 (4.9) | 28.0 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 36

OUTCOME MEASURES:

1. Primary Outcome: Maximum Measured Concentration (Cmax) at Steady State for Telmisartan
Description: Maximum measured concentration (Cmax) of telmisartan in plasma at steady state over the dosing interval tau
Time Frame: 15 minutes (min) before drug administration and 15min, 30min, 45min, 1 hour (h), 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 12h, 24h, 32h, 48h and 72h after 10 days drug administration
Population: Pharmacokinetic (PK) set which included all subjects in the treated set who had evaluable PK variable of test (T80/A5/H12.5 mg) and at least one of two references (T80/H12.5 mg and T80/A5 mg) for treatment periods 1, 2, and 3. Subjects who had a protocol deviation relevant to the evaluation of relative bioavailability were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- T80-A5-H12.5: Participants received oral administration of Telmisartan 80mg/Amlodipine 5mg/HCTZ 12.5mg fixed-dose combination (FDC) tablet (T80-A5-H12.5) once daily for ten days.
- T80-A5: Participants received oral administration of Telmisartan 80mg/Amlodipine 5mg fixed-dose combination tablet (T80-A5) once daily for 10 days
- T80-H12.5: Participants received oral administration Telmisartan 80mg/HCTZ 12.5mg fixed-dose combination tablet (T80-H12.5) once daily for 10 days
Arm/Group | T80-A5-H12.5 | T80-A5 | T80-H12.5
Number analyzed (Participants) | 36 | 34 | 36
ng/mL | 970 (69.3) | 857 (70.7) | 895 (75.0)
Statistical Analysis 1: Comparison: T80-A5-H12.5 vs T80-H12.5; Test type: Non-Inferiority or Equivalence — Non-inferiority limits: 80% - 125%; ANOVA; The model included effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment; Adjusted geometric mean ratio (%) = 108.39, 90% CI 2-sided [93.081 to 126.225], Standard Error of Mean 1.094 — Ratio calculated as T80-A5-H12.5 divided by T80-H12.5
Statistical Analysis 2: Comparison: T80-A5-H12.5 vs T80-A5; Test type: Non-Inferiority or Equivalence — Non-inferiority limits: 80% - 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 114.86, 90% CI 2-sided [98.216 to 134.326], Standard Error of Mean 1.097 — Ratio calculated as T80-A5-H12.5 divided by T80-A5

2. Primary Outcome: Area Under the Plasma Concentration Curve at Steady State for Telmisartan
Description: Area under the plasma concentration curve (AUC) of telmisartan in plasma at steady state over the dosing interval tau
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | T80-A5-H12.5 | T80-A5 | T80-H12.5
Number analyzed (Participants) | 36 | 34 | 36
ng*h/mL | 2510 (72.1) | 2570 (70.8) | 2580 (81.4)
Statistical Analysis 1: Comparison: T80-A5-H12.5 vs T80-H12.5; Test type: Non-Inferiority or Equivalence — Non-inferiority limits: 80% - 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 97.53, 90% CI 2-sided [90.43 to 105.19], Standard Error of Mean 1.05 — Ratio calculated as T80-A5-H12.5 divided by T80-H12.5
Statistical Analysis 2: Comparison: T80-A5-H12.5 vs T80-A5; Test type: Non-Inferiority or Equivalence — Non-inferiority limits: 80% - 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 102.04, 90% CI 2-sided [96.94 to 107.40], Standard Error of Mean 1.03 — Ratio calculated as T80-A5-H12.5 divided by T80-A5

3. Secondary Outcome: Amount of HCTZ Excreted in Urine at Steady State From 0 to 24 Hours
Description: Amount of HCTZ excreted in urine over the time interval from 0 to 24 hours at steady state
Time Frame: 0-6 hours (h), 6-12h and 12-24h after drug administration on day 10
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | T80-A5-H12.5 | T80-H12.5
Number analyzed (Participants) | 36 | 36
mg | 10.4 (11.4) | 9.9 (12.2)
Statistical Analysis 1: Comparison: T80-A5-H12.5 vs T80-H12.5; Test type: Non-Inferiority or Equivalence — Non-inferiority limits: 80% - 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 104.80, 90% CI 2-sided [101.949 to 107.734], Standard Error of Mean 1.016 — Ratio calculated as T80-A5-H12.5 divided by T80-H12.5

4. Primary Outcome: Maximum Measured Concentration (Cmax) at Steady State for Amlodipine
Description: Maximum measured concentration (Cmax) of amlodipine in plasma at steady state over the dosing interval tau
Time Frame: 15 minutes (min) before drug administration and 15min, 30min, 45min, 1 hour (h), 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 12h, 24h, 32h, 48h, 72h, 96h, 120h and 144h after 10 days drug administration
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | T80-A5-H12.5 | T80-A5
Number analyzed (Participants) | 36 | 34
ng/mL | 11.8 (21.8) | 11.3 (22.3)
Statistical Analysis 1: Comparison: T80-A5-H12.5 vs T80-A5; Test type: Non-Inferiority or Equivalence — Non-inferiority limits: 80% - 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 103.95, 90% CI 2-sided [101.023 to 106.964], Standard Error of Mean 1.017 — Ratio calculated as T80-A5-H12.5 divided by T80-A5

5. Primary Outcome: Area Under the Plasma Concentration Curve at Steady State for Amlodipine
Description: Area under the plasma concentration curve (AUC) of amlodipine in plasma at steady state over the dosing interval tau
Time Frame: as for outcome 4
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | T80-A5-H12.5 | T80-A5
Number analyzed (Participants) | 36 | 34
ng*h/mL | 230 (23.4) | 223 (21.8)
Statistical Analysis 1: Comparison: T80-A5-H12.5 vs T80-A5; Test type: Non-Inferiority or Equivalence — Non-inferiority limits: 80% - 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 102.49, 90% CI 2-sided [100.167 to 104.867], Standard Error of Mean 1.014 — Ratio calculated as T80-A5-H12.5 divided by T80-A5

6. Primary Outcome: Maximum Measured Concentration (Cmax) at Steady State for HCTZ
Description: Maximum measured concentration (Cmax) of HCTZ in plasma at steady state over the dosing interval tau
Time Frame: 15 minutes (min) before drug administration and 15min, 30min, 45min, 1 hour (h), 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 12h, 24h, 32h and 48h after 10 days drug administration
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | T80-A5-H12.5 | T80-H12.5
Number analyzed (Participants) | 36 | 36
ng/mL | 107 (28.5) | 102 (28.0)
Statistical Analysis 1: Comparison: T80-A5-H12.5 vs T80-H12.5; Test type: Non-Inferiority or Equivalence — Non-inferiority limits: 80% - 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 105.35, 90% CI 2-sided [99.230 to 111.847], Standard Error of Mean 1.036 — Ratio calculated as T80-A5-H12.5 divided by T80-H12.5

7. Primary Outcome: Area Under the Plasma Concentration Curve at Steady State for HCTZ
Description: Area under the plasma concentration curve (AUC) of HCTZ in plasma at steady state over the dosing interval tau
Time Frame: as for outcome 6
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | T80-A5-H12.5 | T80-H12.5
Number analyzed (Participants) | 36 | 36
ng*h/mL | 584 (23.8) | 565 (23.4)
Statistical Analysis 1: Comparison: T80-A5-H12.5 vs T80-H12.5; Test type: Non-Inferiority or Equivalence — Non-inferiority limits: 80% - 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted geometric mean ratio (%) = 103.39, 90% CI 2-sided [98.730 to 108.280], Standard Error of Mean 1.028 — Ratio calculated as T80-A5-H12.5 divided by T80-H12.5

ADVERSE EVENTS:
Time Frame: 10 days
Groups:
- All Patients: All participants in the study. Participants received three treatments in a randomised order
  * T80-A5-H12.5
  * T80-A5
  * T80-H12.5
Arm/Group | T80-A5-H12.5 | T80-H12.5 | T80-A5 | All Patients
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 3/36 | 3/36 | 2/34 | 5/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T80-A5-H12.5 (N=36) | T80-H12.5 (N=36) | T80-A5 (N=34) | All Patients (N=36)
Alanine aminotransferase increased (Investigations) | 3 | 2 | 2 | 4
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.